CLINICAL TRIAL: NCT00204659
Title: Phase II Study With Rituximab and CHOP in Patients With Gastric Diffuse Large B-Cell Non-Hodgkin's Lymphoma
Brief Title: Phase II Study With Rituximab and Cyclophosphamide, Doxorubicin, Vincristine, Prednisone (CHOP) in Patients With Gastric Diffuse Large B-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Wolfram Brugger, M.D., Schwarzwald-Baar Clinic, Academic Teaching Hospital, Univ. Freiburg
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 64-03
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-09

CONDITIONS: Primary Gastric Diffuse-Large B-Cell Lymphoma
Keywords: Rituximab; CHOP; DLBCL; gastric lymphoma
MeSH Terms: conditions — Familial primary gastric lymphoma | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rituximab + CHOP chemotherapy — standard Rituximab + CHOP chemo-immunotherapy
  Other Names: MabThera

SUMMARY:
The optimal treatment of primary gastric diffuse large B-cell lymphoma (PG-DLBCL) has not yet been defined. In most circumstances, a stomach-conserving approach is favored, but the role of radiotherapy is still a matter of debate. Recently, Rituximab along with full-dose CHOP chemotherapy has been shown to improve the outcome in elderly patients with nodal DLBCL. However, no data are available with such a therapy in patients with PG-DLBCL. Therefore, in March 2003, we initiated an ongoing, prospective, multicenter phase II study in patients with PG-DLBCL with 6 to 8 cycles of Rituximab (R; 375 mg/m2) plus CHOP-21 in order to evaluate the safety and efficacy of this approach.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Histologically confirmed primary gastric CD20+ DLBCL
* Written informed consent
* ECOG 0-2

Exclusion Criteria:

* Secondary aggressive Non-Hodgkin's lymphoma involving the gastric area
* HIV positive patients
* Severe organ dysfunction
* Life expectancy of less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Complete remission rate | at end of chemo-immunotherapy
Progression-free survival | at 2 and 5 years

SECONDARY OUTCOMES:
Overall survival | at 2 and 5 years
Toxicity | after chemo-immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram Brugger, M.D., Principal Investigator — Schwarzwald-Baar Clinic, Academic Teaching Hospital, University of Freiburg
Locations (5):
- Germany (5):
  - Zentralklinikum Augsburg, Augsburg
  - University of Giessen, Giessen
  - Klinikum Reutlingen, Reutlingen
  - University of Tubingen, Tübingen
  - Schwarzwald-Baar Clinic, Villingen-Schwenningen